CLINICAL TRIAL: NCT03178747
Title: A Comparative Study of Tzanck Smear With Methylene Blue Versus Giemsa Stain to Diagnose Herpes Simplex, Herpes Zoster and Varicella Zoster Skin Infections
Brief Title: Tzanck Smear With Methylene Blue Stain for Herpes
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Collaborators: Dermatological Society of Thailand (Other)
Responsible Party: Principal Investigator, Pawinee Rerknimitr, Assistant professor, Chulalongkorn University
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 674/59
Record Dates: First submitted 2017-06-02; First posted 2017-06-07 (Actual); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Herpes Simplex; Herpes Zoster; Varicella Zoster
Keywords: Methylene blue; Giemsa; Tzanck smear
MeSH Terms: conditions — Herpes Simplex; Herpes Zoster

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case (Active Comparator): Patients who clinically diagnosed as herpes simplex, herpes zoster or varicella zoster skin infection.
  Interventions: Diagnostic Test: Methylene blue; Diagnostic Test: Giemsa stain
- Negative control (Sham Comparator): Patients who develops vesicular lesion but not typically considered as herpesviral skin infection, such as acute eczema, Paederus dermatitis
  Interventions: Diagnostic Test: Methylene blue; Diagnostic Test: Giemsa stain

INTERVENTIONS:
Diagnostic Test: Methylene blue — working solution methylene blue
Diagnostic Test: Giemsa stain — working solution Giemsa stain (Wolbach's modification)

SUMMARY:
To compare the sensitivity of Tzanck smear with methylene blue stain versus traditional Giemsa stain in patients with herpes infection.

DETAILED DESCRIPTION:
A smear from the lesional skin of the patients suspected having Herpes simplex, Herpes zoster and Varicella zoster skin infections will be collected (in a clinical routine setting). The specimen will be stained with methylene blue in addition to the Giemsa stain. Polymerase chain reaction study for herpes antigen will be performed in some of the specimens. The sensitivity, specificity, positive predictive value and negative predictive value will be calculated from the results of the study.

ELIGIBILITY:
Inclusion Criteria:

* patients with clinically suspected of having herpes simplex, herpes zoster, varicella zoster skin infections.
* Those who have vesicular skin lesion such as acute eczema, Paederus dermatitis.
* Those are well cooperative.
* Age > 18 years old.

Exclusion Criteria:

* Those who are not willing to have specimen from skin lesions to be collected.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-03-07 (Actual); Primary Completion 2017-12-07 (Estimated); Study Completion 2018-03-06 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | 24 weeks
  Positive results from staining compared with number of cases

SECONDARY OUTCOMES:
Factors that contribute the results from Methylene blue staining | 24 weeks
  Subgroup analysis which included age, sex, clinical morphology, distribution, duration of lesion.
Specificity | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pawinee Rerknimitr, MD, MSc, Principal Investigator — Chulalongkorn University
Locations (1):
- Division of Dermatology, Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No